CLINICAL TRIAL: NCT04797923
Title: A Phase II Study Evaluating Efficacy and Safety of Conversion Surgery After Intraperitoneal Paclitaxel in Combination With Systemic Capecitabine and Oxaliplatin Chemotherapy in Advanced Gastric Cancer Patients With Peritoneal Dissemination
Brief Title: A Phase II Study of Conversion Surgery After IP Paclitaxel With XELOX Chemotherapy in AGC With Peritoneal Dissemination
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Seung Ho Choi, Professor, Gangnam Severance Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3-2020-0237
Record Dates: First submitted 2021-03-11; First posted 2021-03-15 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Advanced Gastric Cancer; Peritoneal Carcinomatosis
Keywords: Intraperitoneal chemotherapy, Conversion surgery, Advanced gastric cancer, peritoneal carcinomatosis
MeSH Terms: conditions — Peritoneal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intraperitoneal paclitaxel with systemic chemotherapy (Experimental)
  Interventions: Drug: 1. Treatment: IP chemotherapy + Systemic chemotherapy; Procedure: 2. Response evaluation after 4 cycles of IP + systemic chemotherapy

INTERVENTIONS:
Drug: 1. Treatment: IP chemotherapy + Systemic chemotherapy — 1. Treatment: IP chemotherapy + Systemic chemotherapy Day1 + Day 8: IP Paclitaxel 40 mg/m2 every 3 weeks Day1: IV Oxaliplatin 100 mg/m2 every 3 weeks Day 1~14: Capecitabine 1000 mg/m2 PO, BID every 3 weeks
Procedure: 2. Response evaluation after 4 cycles of IP + systemic chemotherapy — 2. Response evaluation after 4 cycles of IP + systemic chemotherapy
  * Conversion surgery will be done following diagnostic laparoscopy after 4 cycles of IP + systemic chemotherapy. Additional 4 cycles of IP + systemic chemotherapy wille be done following surgery.
  * If surgery is impossible after 4th cycle, four additional cycles of treatment will be done, and convertibility will be evaluated.
  * IP chemotherapy should not exceed total of 8 cycles.

SUMMARY:
Advanced gastric cancer combined with peritoneal seeind has dismal prognosis with poor response to systemic chemotherapy and with rapid aggravation of symptoms such as abdominal pain, ileus, and poor nutritional intake. Intraperitoneal (IP) chemotherapy through IP port or catheter has lower complication than HIPEC (hyperthermic intraperitoneal chemotherapy) and can deliver higher dose of chemotherapy with less systemic toxicity. IP chemotherapy combined with systemic chemotehrapy showed benefit in several clinical trials, despite lack of statistical significance in phase 3 clinical trial. Proper dose/combination of chemotherapeutic agents and indication of IP chemotherapy should be investigated through prospective, large-scale clinical trials.

Conversion surgery after cytotoxic chemotherapy showed improved survival in retrospective studies. Our hypothesis is that IP chemotherapy combined with systemic chemotherpay (capecitabine + oxaliplatin) would improve success rate of conversion surgery with R0 resection. In the present study, the treatment regimen consists of intraperitoneal paclitaxel combined with oxaliplatin and capecitabine (XELOX), and will be performed following surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed advanced gastric cancer adenocarcinoma
2. Peritoneal metastasis histopathologically confirmed by laparoscopy or laparotomy and PCI <12 (including patients with no gross peritoneal lesion and cytology positive)
3. No prior surgery for curative aim and previous chemotherapy for recurrent/metastatic gastric cancer
4. Patient who is willing and able to provide written informed consent/assent for the trial
5. Age between 19 and 75 years
6. Measurable lesion according to RECIST 1.1 criteria
7. ECOG performance status 0-1
8. Have adequate organ function

   * ANC ≥ 2,000/uL,
   * hemoglobin ≥ 9.0g/dL
   * platelet ≥ 100,000/uL
   * total Bilirubin: ≤ 1.5 × upper normal limit
   * Creatinine ≤ 1.5 × upper normal limit or Creatinine clearance ≥ 60ml/min
   * AST/ALT ≤ 3.0 x upper normal limit
   * Albumin ≥ 2.5 g/dL
   * PT or INR, aPTT ≤ 1.5 × upper normal limit
9. Should agree to use an adequate method of contraception

Exclusion Criteria:

1. Previous systemic chemotherapy for metastatic/recurrent advanced gastric cancer
2. Patient who has distant metastasis or para-aortic lymph node metastasis or retroperitoneal metastasis except peritoneal metastasis. (But the patient who has ovarian metastasis with resectable status can be enrolled.)
3. Primary tumor cannot be resected because of direct invasion to other important organ. (But, if the invaded organ can be resected together, such as spleen, gallbladder, distal pancreas, and liver, the patient can be enrolled)
4. BMI ≤ 18.5 kg/m2
5. HER2 positive patient (IHC 3+, 2+ with in situ hybridization +)
6. Remnant gastric cancer
7. Intolerable to oral intake of chemotherapeutic agent or have malabsorption syndrome
8. Known additional malignancy that is progressing or requires active treatment in recent 3 years (excluding skin basal cell carcinoma, skin squamous cell carcinoma, thyroid cancer, or in situ cervix cancer that has undergone potentially curative therapy)
9. Symtomatic CNS metastasis and/or leptomeningeal seeding
10. Autoimmune disease in recent 2 years requiring systemic therapy
11. Clinically significant heart disease
12. Peripheral neuropathy ≥ Grade 2
13. Pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment
14. History of HIV, HBV, or HCV

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Rate of R0 resection | 30 days after the surgery
  Success rate of conversion surgery (Rate of R0 resection)

CONTACTS AND LOCATIONS:
Locations (1):
- Gangnam Severacne Hospital, Seoul, Gangnnam, South Korea